CLINICAL TRIAL: NCT02503592
Title: Vestibular Function After Cochlear Implantation Using Soft Surgery Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00060216
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Vestibular Function in Cochlear Implant Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cochlear Implant group - Vestibular testing (Active Comparator): Adult patients who have been implanted with a Med-El Cochlear implant device within the last 3 months who completed pre-op vestibular testing as standard of care. These subjects will undergo a series of post-op vestibular testing, at the 3 month and 12 month follow up visits
  Interventions: Other: Vestibular testing
- Control Group - existing historical vestibular data (No Intervention): This group will consist of existing historical vestibular testing data only. No subjects will be enrolled on this arm.

INTERVENTIONS:
Other: Vestibular testing — Patients who have received a cochlear implant within 90 days, and had vestibular testing pre-operatively, will undergo post-op vestibular testing
  Arms: Cochlear Implant group - Vestibular testing

SUMMARY:
This study will measure the effects of soft surgical techniques on vestibular function and quality of life in patients pre- and post-cochlear implant (CI) surgery. Additionally, the investigators will attempt to systematically evaluate the utility of different electrophysiological measures of vestibular system function in surgical ears.

Vestibular system function in CI patients will be evaluated pre-surgically and twice post-surgically, at 3 months and again at 1 year post-surgery. Traditional test techniques - such as VNG, rotational testing, and air conduction VEMPs - will be compared to and cross-checked with newer techniques including video head impulse testing (vHIT) and bone conduction VEMPs.

DETAILED DESCRIPTION:
Design & Procedures: The current standard of care for CI patients includes a pre-op evaluation of the vestibular system. For this study, the investigators will compare subjects' routine pre-op test results to two additional post-op assessments performed for study purposes: one in the short term (~3 months post-op) and one in the long-term (~1 year post-op).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Only patients implanted with the MED-EL CI device within the last 90 days will be eligible for this study.

Exclusion Criteria:

* Patients < 18 years of age
* Patients implanted with a cochlear implant device other than MED-El CI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04; Primary Completion 2018-05-30 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Vestibular function in Cochlear Implant Patients | Pre-Operatively, and then 3 months and 12 months post-operatively
  Vestibular system function in CI patients will be evaluated pre-surgically and twice post-surgically, at 3 months and again at 1 year post-surgery
Change in Quality of Life by questionnaire | 3 months and 12 months post-operatively
  Self-reported quality of life questionnaire (DHI) will be collected 3 months and 12 months post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Piker, AuD, PhD,, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States